CLINICAL TRIAL: NCT07059572
Title: Comparative Evaluation of Guava Leaf Extract and Chlorhexidine Mouthwash in Patients With Chronic Gingivitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Shakila Jahan Nabila, Principal investigator, MD, Dental Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5516
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Gingivitis, Plaque Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B-0.2% Chlorhexidine mouthwash group (Active Comparator): Participants will be instructed to rinse with 10 ml of 0.2% Chlorhexidine Mouthwash twice daily for 30 and 90 days. Each rinse will last for 1 minute, after which the mouthwash is to be expectorated without swallowing.
  Interventions: Drug: Group B- 0.2% Chlorhexidine mouthwash
- Group A- 0.15% Guava Leaf Extract Mouthwash (Experimental): Participants will be instructed to rinse with 10 ml of 0.15% Guava Leaf Extract Mouthwash twice daily for 30 and 90 days. Each rinse will last for 1 minute, after which the mouthwash is to be expectorated without swallowing.
  Interventions: Drug: Group A- 0.15% Guava leaf extract mouthwash group

INTERVENTIONS:
Drug: Group A- 0.15% Guava leaf extract mouthwash group — Participants will be instructed to rinse with 10 ml of 0.15% Guava Leaf Extract Mouthwash twice daily for 30 and 90 days. Each rinse will last for 1 minute, after which the mouthwash is to be expectorated without swallowing.
  Arms: Group A- 0.15% Guava Leaf Extract Mouthwash
Drug: Group B- 0.2% Chlorhexidine mouthwash — Participants will be instructed to rinse with 10 ml of 0.2% Chlorhexidine Mouthwash twice daily for 30 and 90 days. Each rinse will last for 1 minute, after which the mouthwash is to be expectorated without swallowing."
  Arms: Group B-0.2% Chlorhexidine mouthwash group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of 0.15% guava (Psidium guajava) leaf extract mouth rinse with 0.2% Chlorhexidine (CHX) mouth rinse in reducing plaque accumulation, gingival inflammation, and oral microbial load in participants with plaque-induced chronic moderate or severe gingivitis. Half of the participants will receive guava leaf extract mouth rinse, and the other half will receive Chlorhexidine(CHX).

DETAILED DESCRIPTION:
Plaque-induced gingivitis is one of the most prevalent oral health problems worldwide and, if not addressed, can progress to periodontitis with irreversible loss of supporting tissues. Although mechanical plaque control through tooth-brushing and flossing is essential, many individuals do not achieve adequate plaque removal, so antimicrobial mouth rinses are commonly prescribed as adjuncts. The standard 0.2 % chlorhexidine (CHX) rinse is effective yet limited by tooth staining, taste alteration, and mucosal irritation, prompting interest in safer natural options. Psidium guajava (guava) leaf extract contains flavonoids, tannins, and other bioactive compounds with documented antimicrobial, anti-inflammatory, and antioxidant properties and has shown promise as a natural oral-care agent. This clinical trial will be conducted in the Out-patient Department and will enrol 160 adults with plaque-induced chronic moderate or severe gingivitis selected by purposive sampling method. After baseline non-surgical periodontal therapy, participants will be allocated to an intervention group that receives a 0.15 % guava-leaf extract mouth rinse or to a control group that receives a 0.2 % Chlorhexidine(CHX) mouth rinse; each participant will rinse with 10 mL twice daily, 30 minutes after brushing, for three months. Plaque Index (Turesky modification of Quigley-Hein) and Gingival Index (Löe & Silness) will be recorded at baseline, one month, and three months to gauge changes in plaque accumulation and gingival inflammation. To explore antimicrobial performance, the study will determine zones of inhibition and minimum inhibitory concentration (MIC) values for each rinse. Participants will also complete structured questionnaires on taste, staining, burning sensation, and overall acceptability, and any adverse events will be documented. Findings from this trial will clarify whether guava-leaf mouth rinse offers clinical and antimicrobial benefits comparable to, or better than, Chlorhexidine(CHX) while avoiding its common side-effects, potentially providing a locally sourced, culturally acceptable, and affordable adjunct for managing gingivitis in Bangladesh and similar settings.

ELIGIBILITY:
Inclusion Criteria: • Participants with a minimum of 24 functional teeth.

* Presence of Plaque induced chronic moderate to severe form of gingivitis.
* Participants within the age group of 18 to 35 years.
* Willing and able to comply with all study procedures.

Exclusion Criteria: • Pregnant or lactating women.

* Systemically compromised people; subjects with removable or fixed orthodontic appliances or prosthesis.
* People who were prescribed antibiotics or inflammatory drugs in the past 1 month.
* History of smoking or any form of tobacco use.
* History of allergic reactions to Chlorhexidine or Guava.
* Severe systemic conditions that could contraindicate participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Plaque Index | At baseline, 1 month, and 3 months post-intervention
  Plaque Index (PI) will be assessed using the Turesky-Gilmore-Glickman modification of the Quigley-Hein index. This index measures the extent of dental plaque accumulation on six surfaces per tooth and assigns scores from 0 (no plaque) to 5 (plaque covering more than two-thirds of the surface). The average PI score will be calculated for each participant and compared over time to determine the plaque-reducing efficacy of guava leaf extract versus 0.2% chlorhexidine.
Change in Gingival Index (GI) | At Baseline, 1 Month, and 3 Months post-intervention
  Gingival Index (GI) will be used to assess the degree of gingival inflammation. It will be measured using the Löe and Silness index, which scores each gingival unit (mesial, distal, buccal, and lingual) on a scale from 0 to 3. A score of 0 indicates normal gingiva, while 3 indicates severe inflammation with marked redness, edema, ulceration, and spontaneous bleeding. The mean GI score will be compared across the three time points to evaluate the anti-inflammatory effects of guava leaf extract versus 0.2% chlorhexidine mouthwash.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Dhaka Division, Bangladesh